CLINICAL TRIAL: NCT05684653
Title: An Open-Label, Parallel, Single-dose, Phase I Clinical Study to Evaluate the Pharmacokinetics and Safety of Orelabrutinib Tablets in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: Study to Evaluate Orelabrutinib Tablets in Subjects With Hepatic Impairment and Healthy Subject
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICP-CL-00119
Record Dates: First submitted 2022-12-14; First posted 2023-01-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib Tablets (Experimental): Subjects take Single dose of 50 mg orelabrutinib tablet under fasting state
  Interventions: Drug: Orelabrutinib Tablets

INTERVENTIONS:
Drug: Orelabrutinib Tablets — 50 mg, single oral dose

SUMMARY:
This is an Open-Label, Parallel, Single-dose, Phase I Clinical Study to Evaluate the Pharmacokinetics and Safety of Orelabrutinib Tablets in Subjects with Varying Degrees of Hepatic Impairment

ELIGIBILITY:
Inclusion Criteria:

1. The subject understands and has provided the informed consent form (ICF);
2. Male and female between 18 and 79 years old (inclusive) at the time of signing the ICF;
3. Male with weight not less than 50 kg and female not less than 45 kg. Body mass index (BMI): 18-32 kg/m2 (inclusive);
4. The subject is suitable to participate in the study as evaluated by the investigator based on physical examination, vital signs, laboratory tests, and 12-lead ECG;
5. Within 2 weeks before the study medication, the subject took no prohibited drug (see Appendix 4 for the contraindicated drugs), including any prescription drug, OTC drug, Chinese herbal medicine, or dietary supplement;
6. The subject is willing to take effective contraception voluntarily from the screening to 3 months after the dosing of study drug;

The following criteria apply to the subjects with hepatic impairment:

Patients with chronic hepatic impairment resulted from viral hepatitis, alcoholic liver disease, autoimmune hepatitis, or other causes. Patients with chronic hepatic impairment are defined as patients with a history of hepatic impairment and stable liver functions for ≥ 1 month based on clinical manifestations. For patients with viral hepatitis, it is imperative to exclude active hepatitis C (if the patient was tested HCV antibody positive, at least 2 tests within 3 months indicating HCV-RNA negative are required) and active hepatitis B (HBV-DNA level should be less than 100 IU/mL with concurrent antiviral treatment); or patients with hepatic cirrhosis confirmed by liver biopsy or other medical imaging (including laparoscopy, computed tomography (CT), magnetic resonance imaging (MRI), or ultrasonography); or patients with diagnosed hepatic cirrhosis complicated with portal hypertension (allow receiving related portal hypotensives treatments, e.g., carvedilol). Patients who meet any of the above conditions can participate in this study.

8. Hepatic impairment of Class A or Class B or Class C based on Child-Pugh system (no albumin should be used within 14 days); and resulted from prior primary liver disease; 9. Coagulation functions: INR≤2.5 without intervention of coagulants (2-week washout); hematology: neutrophil count ≥ 1.5 × 109/L, hemoglobin ≥ 70 g/L, platelet count ≥30 × 109/L; hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × upper limit of normal (ULN); 10. Stable therapy for hepatic impairment before the study medication, and at least 4-week stable medication for treatment of hepatic impairment (stable medications were judged by the investigator); 11. The subject agrees to abstain from smoking, alcohol, caffeinated beverages, and fruit juice beverages from 7 days before the study medication to the end of study follow-up.

Exclusion Criteria:

1. Drug-induced liver injury;
2. Acute hepatic impairment due to various causes;
3. Any of the following circumstances: liver transplant recipients; acute or exacerbating hepatic impairment due to various causes; liver failure, complicated with grade 3/4 hepatic encephalopathy; active lesions of hepatic cancer; esophageal and gastric varices hemorrhage; serious/advanced peritoneal or pleural effusion requiring puncture drainage and albumin supplementation; situations deemed not suitable to participate in the study including hepatorenal syndrome;
4. Diseases influencing bile excretion within 3 months before the screening, including cholestatic liver disease or biliary tract infection;
5. Subjects having portal hypertension with esophageal and gastric varices bleeding within 3 months or subjects having received portal-systemic shunt procedure within half a year, including transjugular intrahepatic portosystemic shunt (TIPS);
6. History of significant allergy or intolerance to any drug, food, or other substance;
7. Patients with abnormal test value which is clinical significance at screening or before enrollment, that influence the evaluation of safety, including physical examination, vital signs, routine laboratory tests (hematology, blood biochemistry, coagulation function, and urinalysis), 12-lead ECG, and chest CT;
8. Any history of serious disease or tother conditions that may influence the study findings, including but not limited to disorders of nervous, cardiovascular, hematologic and lymphatic, immune, renal, gastrointestinal, respiratory, endocrine systems;
9. History of surgery that may influence drug absorption, distribution, metabolism, or excretion (e.g., gastroduodenectomy), or proposed possible surgery or scheduled hospitalization during the study;
10. Clinical manifestations of bacterial, viral, parasitic, or fungal infection requiring treatment, and coronavirus infection or nucleic acid test positive at screening (excluding hepatitis B) or history of serious active infection within 1 month before the screening;
11. Human immune-deficiency virus (HIV) antibody positive or active syphilis at screening;
12. Anticoagulation therapies including warfarin or thrombin inhibitors and/or antiplatelet therapy with aspirin within 1 month before the screening;
13. Administration of inhibitors or inducers of drug metabolism in the liver, administration of sensitive P-gp and BCRP substrates with narrow therapeutic index within 2 weeks (or 5 half-lives, whichever longer) before the screening;
14. Drug abuse or history of soft drugs within 3 months before the screening or history of hard drugs within 1 year before the screening; or urine drug test positive at screening;
15. Mean daily consumption of more than 5 cigarettes or habitually consumption of nicotine-containing products , mean daily alcohol intake exceeds the criteria within 3 months before the screening with failure to abstain from smoking or or cannot abstain from alcohol during the trial;
16. Intake of grapefruit juice, methylxanthine-rich food or beverages (e.g., coffee, tea, cola, chocolates, and energy drinks) within 7 days before taking the study medication, or strenuous exercise or any other factor influencing drug absorption, distribution, metabolism, and excretion, with failure to abstain from during the trial;
17. Those who participated in clinical trials of any other study drug or medical device within 3 months before the first dose of the study drug, or participated in 3 or more clinical trials of drugs or medical devices within the latest year; for other study drugs with a long half-life, a longer time interval is required for at least 5 half-lives of the drug;
18. Blood donation (or lost) ≥ 400 mL within 3 months before the screening, or blood transfusion recipients or blood product users;
19. Vaccination within 4 weeks before the screening or scheduled vaccination during the trial;
20. Women in lactation or with serum pregnancy test positive at screening;
21. Birth plan scheduled from screening to 3 months after trial completion, or unwilling to take rigorous contraception from screening to 3 months after study completion, or proposed scheduled sperm donation;
22. Unwilling or Unable to abide by the study procedure specified in the protocol, or has any factor deemed unsuitable for participating in this clinical study by the investigator.

    The following exclusion criteria apply to subjects with normal hepatic function:
23. History of hepatic impairment, or presence of possible hepatic impairment at screening as suggested by physical examination and laboratory tests; HBsAg-positive or anti-HCV antibody-positive.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Area under the concentration-time curve from time 0 to infinity (AUC0-t) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose , at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Maximum concentration(Cmax) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.

SECONDARY OUTCOMES:
Time to maximum concentration（Tmax）(Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Half-Life (T1/2) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Apparent Volume of Distribution (Vz/F) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Apparent clearance (CL/F) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Unbound maximum concentration (Cmax, unb) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose.
Area under the unbound drug concentration-time curve (AUCunb) (Blood) | Blood samples for pharmacokinetics will be taken on Day 1 at pre dose, at 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48hours post dose.
AEs | Through study completion, an average of 1 year
SAEs | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affilitaed Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affilitaed Hospital of Soochow University, Suzhou, Jiangsu
  - Deyang People's Hospital, Deyang, Sichuan
  - Shulan (Hangzhou) hospital, Hangzhou, Zhejiang